CLINICAL TRIAL: NCT06958146
Title: Impact of Single Dose Azithromycin During Labor on Maternal and Neonatal Infections
Brief Title: Azithromycin for Preventing Maternal and Neonatal Infections During Labor.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, professor, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Azithromycin 2025
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Maternal and Neonatal Sepsis; Intrapartum Antibiotics
MeSH Terms: conditions — Neonatal Sepsis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregnanct ladies in labor receiving single dose azithromycin along with standard labor care (Experimental): The participants in this arm will receive a single dose of 2 g oral azithromycin along with standard care in the intrapartum period
  Interventions: Drug: oral azithromycin
- Pregnant ladies in labor receiving only standard care and no oral azithromycin (Placebo Comparator): participants in this arm will be given only standard labor care and no antibiotics
  Interventions: Other: no azithromycin

INTERVENTIONS:
Drug: oral azithromycin — we will be administering single-dose oral azithromycin to ladies who go into labor and have no risk factors for sepsis, as there is increased risk of postpartum sepsis in both mother and neonate after normal vaginal delivery in low-income and middle-income countries
  Arms: pregnanct ladies in labor receiving single dose azithromycin along with standard labor care
Other: no azithromycin — participants in this arm will be given only standard labor care and no oral azithromycin
  Arms: Pregnant ladies in labor receiving only standard care and no oral azithromycin

SUMMARY:
In this study, we want to see the role of the antibiotic, azithromycin, in preventing maternal and neonatal infections, if the drug is given intrapartum to the mother

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies with no risk factors for sepsis who go into spontaneous labor or induced labor

Exclusion Criteria:

* pregnant with risk factors for sepsis like maternal fever , raised WBC count, chorioamnionitis, or having. history of any adverse even with macrolides

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
maternal infections | birth to 6 weeks post partum

SECONDARY OUTCOMES:
neonatal infections | birth to 6 weeks post partum

IPD SHARING:
Plan to Share IPD: Yes
we will upload the data on the website on clinicaltrials.gov
Supporting Information: Study Protocol